CLINICAL TRIAL: NCT03635788
Title: A Phase III Study to Evaluate Long-Acting Antiretroviral Therapy in Non-Adherent HIV-Infected Individuals
Brief Title: The LATITUDE Study: Long-Acting Therapy to Improve Treatment SUccess in Daily LifE
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: ViiV Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACTG A5359; 30104 (Registry Identifier: DAIDS-ES Registry Number)
Record Dates: First submitted 2018-08-15; First posted 2018-08-17 (Actual); Results first posted 2025-04-24 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-04

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — Standard of Care; Rilpivirine; cabotegravir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Step 1 SOC (Other): In Step 1, participants received SOC oral ART regimen for up to 24 weeks.
  Interventions: Drug: Standard of Care (SOC) Oral ART
- Step 2 Arm A: LA ART (Experimental): In Step 2, participants received oral RPV once daily and oral CAB once daily for 4 weeks (optional), followed by a RPV-LA loading dose and a CAB-LA loading dose, followed in 4 weeks by an RPV-LA maintenance dose and a CAB-LA maintenance dose every 4 weeks for 44 weeks.
  Interventions: Drug: Oral RPV; Drug: Oral CAB; Drug: RPV-LA Loading Dose; Drug: CAB-LA Loading Dose; Drug: RPV-LA Maintenance Dose; Drug: CAB-LA Maintenance Dose
- Step 2 Arm B: SOC (Active Comparator): In Step 2, participants continued SOC oral ART regimen for 52 weeks.
  Interventions: Drug: Standard of Care (SOC) Oral ART

INTERVENTIONS:
Drug: Standard of Care (SOC) Oral ART — SOC oral ART regimen must include at least 3 drugs with 2 or more drugs predicted to be fully active, including a boosted protease inhibitor (PI) and/or an integrase strand transfer inhibitor (INSTI)
  Arms: Step 1 SOC; Step 2 Arm B: SOC
Drug: Oral RPV — RPV 25 mg tablets
  Other Names: Rilpivirine
  Arms: Step 2 Arm A: LA ART
Drug: Oral CAB — CAB 30 mg tablets
  Other Names: Cabotegravir; GSK1265744
  Arms: Step 2 Arm A: LA ART
Drug: RPV-LA Loading Dose — 900 mg administered as one 3 mL (900 mg) intramuscular injection in the gluteal muscle
  Other Names: Rilpivirine Long-Acting Injectable
  Arms: Step 2 Arm A: LA ART
Drug: CAB-LA Loading Dose — 600 mg administered as one 3 mL (600 mg) intramuscular injection in the gluteal muscle
  Other Names: Cabotegravir Long-Acting Injectable
  Arms: Step 2 Arm A: LA ART
Drug: RPV-LA Maintenance Dose — 600 mg administered as one 2 mL (600 mg) intramuscular injection in the gluteal muscle
  Other Names: Rilpivirine Long-Acting Injectable
  Arms: Step 2 Arm A: LA ART
Drug: CAB-LA Maintenance Dose — 400 mg administered as one 2 mL (400 mg) intramuscular injection in the gluteal muscle
  Other Names: Cabotegravir Long-Acting Injectable
  Arms: Step 2 Arm A: LA ART

SUMMARY:
The purpose of this study was to compare the efficacy, safety, and durability of two different strategies to treat participants with a history of sub-optimal adherence and control of their HIV infection: long-acting (LA) antiretroviral therapy (ART) and all-oral standard of care (SOC).

DETAILED DESCRIPTION:
This study compared the efficacy, safety, and durability of two different strategies to treat participants with a history of sub-optimal adherence and control of their HIV infection: long-acting (LA) antiretroviral therapy (ART) with rilpivirine (RPV) LA and cabotegravir (CAB) LA versus all-oral standard of care (SOC).

As the study was originally designed, the study included four steps.

Step 1, Induction

Previously non-adherent individuals were enrolled and underwent a period (up to 24 weeks) of induction SOC ART regimen using conditional economic incentives (CEI). Participants who achieved virologic suppression criteria at or after Step 1, week 4, defined as: a) HIV-1 RNA ≤200 copies/mL or b) HIV-1 RNA of 201-399 copies/mL followed by HIV-1 RNA ≤200 copies/mL by Step 1, week 24, were eligible to enter Step 2.

Step 2, Randomization

Eligible participants were randomized at Step 2 entry in a 1:1 ratio to either of the two treatment arms:

Arm A (LA ART): A combination of oral RPV + oral CAB for 4 weeks (optional) followed by the LA ART Phase, consisting of a two-drug regimen using RPV-LA + CAB-LA Q4 weeks until the end of Step 2 (Table 5.2.1-2). The option to initiate LA ART at the Step 2 Randomization visit without oral RPV + oral CAB was at the discretion of the site investigator of Record (IoR) and participant (see section 2.1, Direct-to-Inject).

Arm B (SOC): Continuation of the SOC for 52 weeks.

Step 3, Continuation/Crossover

Arm A participants continued on RPV-LA + CAB-LA Q4 weeks for 52 weeks until the end of Step 3. Arm B participants (continuation of SOC) who achieved virologic suppression (HIV-1 RNA ≤200 copies/mL) at Step 2, week 48, or HIV-1 RNA of 201-399 copies/mL at Step 2, week 48, followed by HIV-1 RNA ≤200 copies/mL by Step 2, week 52, had the option to cross over at the end of Step 2 to oral RPV + oral CAB for 4 weeks (optional) followed by RPV-LA + CAB-LA every 4 weeks until the end of Step 3 (Table 5.2.1-3). Arm B participants who did not wish or were not eligible to cross over completed study follow-up at Step 2, week 52.

If RPV-LA + CAB-LA became available before a participant finished Step 3, and the participant chose to continue RPV-LA + CAB-LA as part of their clinical care, their follow-up in the study ended at the completion of Step 3. If for some reason the participant chose not to continue LA ART at the end of Step 3 or if LA ART was not available, the participant registered to Step 4 and was followed on locally sourced oral ARV for 52 weeks.

Step 4, Observation

Participants who registered to Step 4 were followed for up to 52 weeks on oral ART. In addition, any participant who received at least one dose of CAB-LA or RPV-LA at any step, and prematurely discontinued the LA ART prior to the end of Step 3, completed their respective Step (either Step 2 or 3) on study/off study treatment, and registered to Step 4 and were followed to complete 52 weeks total on oral ART after their last dose of any LA injectable.

If LA ART became available during follow-up in Step 4, and the participant and provider decided to restart LA ART, they were allowed to do so. In that case, the participants were not followed by the study after restarting LA ART.

On February 12, 2024, based on the interim efficacy results, Data Safety and Monitoring Board (DSMB) recommended stopping randomization to Step 2 and transitioning all eligible participants in Steps 1 and 2 to LA-ART. Per recommendations from DSMB, randomization into Step 2 stopped on February 16, 2024, leaving three steps in the current study protocol 4.0:

In Step 1, participants will receive a SOC oral induction regimen consisting of an ART regimen that involves at least 3 drugs for 24 weeks. Participants who achieve milestones will receive conditional economic incentives. With randomization into Step 2 ended, all eligible Step 1 participants will register to Step 3 at the completion of Step 1.

Participants who are currently on Step 2:

Eligible participants in Step 2 Arm A (already on RPV-LA + CAB-LA) will register to Step 3 and continue on this regimen until the end of Step 3 (52 weeks; See protocol for more information). This should happen at the next scheduled study visit after approval of Version 4.0.

Eligible participants in Step 2 Arm B (SOC arm) will register to Step 3 and switch to oral RPV + oral CAB for 4 weeks (optional; see protocol for more information) followed by RPV-LA + CAB-LA Q4 weeks until the end of Step 3 (52 weeks). This should happen at the next scheduled study visit after approval of Version 4.0.

Eligible participants will enter Step 4 and be followed up to 52 weeks on locally sourced oral ART.

Participants will be followed for up to a total of 180 weeks. Study visits, which will occur throughout the study, may include physical examinations; blood, urine, and hair collection; liver function tests; questionnaires; and an electrocardiogram (ECG).

NOTE: Data summarized in the primary analysis report were based on evaluations undertaken at visits conducted prior to the implementation of Protocol v4.0 which incorporated February 12, 2024 DSMB recommendations. Primary analyses were outlined in the A5359 primary Statistical Analysis Plan (SAP) version 6.0 (dated August 5, 2024) focusing on follow-up in Step 1 and Step 2.

ELIGIBILITY:
Step 1 Inclusion Criteria

HIV-1 infection, documented by any licensed rapid HIV test or HIV enzyme or chemiluminescence immunoassay (E/CIA) test kit at any time prior to study entry and confirmed by a licensed Western blot or a second antibody test by a method other than the initial rapid HIV and/or E/CIA, or by HIV-1 antigen, plasma HIV-1 RNA viral load.

NOTE: The term "licensed" referred to an FDA-approved kit, which was required for all IND studies.

WHO (World Health Organization) and CDC (Centers for Disease Control and Prevention) guidelines mandated that confirmation of the initial test result had to use a test that was different from the one used for the initial assessment. A reactive initial rapid test had to be confirmed by either another type of rapid assay or an E/CIA that was based on a different antigen preparation and/or different test principle (e.g., indirect versus competitive), or a Western blot or a plasma HIV-1 RNA viral load.

HIV-1 Plasma viral load (VL) greater than 200 copies/mL within 12 months prior to study entry by any US laboratory that had a Clinical Laboratory Improvement Amendments (CLIA) certification or its equivalent, unless the participant had been lost to clinical follow-up (see protocol for more information) and no viral load result was available within the last 12 months.

NOTE: Participants who satisfied non-adherence eligibility due to loss to clinical follow-up might not have had a viral load result available at the time of consideration for eligibility. Those participants could be screened and, regardless of their screening viral load result (either ≤ or >200 copies/mL), they would have been eligible for study entry if they met all other inclusion/exclusion criteria.

Evidence of non-adherence to ART according to at least one of the following criteria:

Poor virologic response within 18 months prior to study entry (defined as less than 1 log10 decrease in HIV-1 RNA or HIV-1 RNA greater than 200 copies/mL at two time points at least 4 weeks apart) in individuals who had been prescribed ART for at least 6 consecutive months.

Lost to clinical follow-up within 18 months prior to study entry with ART non-adherence for greater than or equal to 6 consecutive months.

NOTE: Lost to clinical follow-up was defined as either no contact with the provider or missing greater than or equal to 1 appointment in a 6-month period. ART non-adherence was defined as a lapse in ART greater than or equal to 7 days (consecutive or non-consecutive), in the 6-month period where they were lost to clinical follow-up per participant report.

No evidence of any clinically relevant RPV or INSTI resistance-associated mutations (see protocol for more information) through commercially available genotypic (or phenotypic, if available) analyses from any laboratory that had a CLIA certification or equivalent within 60 days of study entry (see protocol for more information), nor history of such mutations on review of prior HIV-1 drug resistance tests by the site investigator. For participants in whom a screening HIV-1 conventional genotype could not be resulted by the testing laboratory, review of historical genotypes and treatment history by the IoR could be used to satisfy this criterion as indicated in the protocol.

Ability of site clinician, in conjunction with the participant, to construct an oral induction antiretroviral (ARV) regimen that had to include at least three ARVs of which at least two had to be predicted to be fully active. The regimen had to include PI/cobi and/or an INSTI based on screening and/or historic resistance testing.

Laboratory values obtained within 60 days prior to study entry by any laboratory that had a CLIA certification or its equivalent:

Hemoglobin greater than or equal to 9.0 g/dL

Absolute neutrophil count (ANC) greater than or equal to 600/mm^3

Alanine aminotransferase (ALT) less than or equal to 3 x upper limit of normal (ULN)

Creatinine Clearance (CrCl) greater than or equal to 50 mL/min estimated by Chronic Kidney Disease Epidemiology Collaboration equation (CKD-Epi).

For participants of reproductive potential, a negative serum or urine pregnancy test with a sensitivity of less than or equal to 25 mIU/mL at screening. This was repeated again at study entry.

NOTE: Participants were considered to be NOT of reproductive potential if: 1) they had had amenorrhea for at least 12 consecutive months prior to study entry (i.e., who had had no menses within 12 months prior to study entry), and had a documented follicle-stimulating hormone (FSH) greater than 40 IU/mL; OR 2) an FSH level was not available, but they had had 24 consecutive months of amenorrhea (in the absence of medications known to induce amenorrhea); OR 3) they reported having undergone surgical sterilization (e.g., hysterectomy, or bilateral oophorectomy, or bilateral tubal ligation/hysteroscopic tubal occlusion).

Contraception Requirements

Participants of Reproductive Potential: Participants of reproductive potential, who were participating in sexual activity that could lead to pregnancy, had to agree to use at least one of the listed highly effective methods for contraception from 30 days prior to the first dose of study medication, while receiving the study drugs, and for 30 days after stopping oral medications, or the duration specified in the product label if receiving study drugs not supplied by the study, or 52 weeks after stopping RPV-LA or CAB-LA. Acceptable methods of contraception included:

Contraceptive subdermal implant

Intrauterine device or intrauterine system

Combined estrogen and progestogen oral contraceptive

Injectable progestogen

Contraceptive vaginal ring

Percutaneous contraceptive patches

Participants Who Were Not of Reproductive Potential: Participants who were not of reproductive potential were eligible to start study drugs without requiring the use of contraceptives. Any statement of self-reported sterility or that of her partner's had to be entered in the source documents.

NOTE A: Acceptable documentation of lack of reproductive potential was the participant's self-reported history of surgical sterilization, menopause, or male partner's azoospermia.

NOTE B: ALL participants in the study were to be counseled on safer sexual practices including the use and benefit/risk of effective barrier methods (e.g., male condom) and on the risk of HIV transmission to a partner without HIV.

Ability and willingness of participant or legal guardian/representative to provide written informed consent.

Step 1 Exclusion Criteria

Currently pregnant, planning to become pregnant during the study period, or currently breastfeeding.

Participants determined by the Site Investigator to have had a high risk of seizures, including participants with an unstable or poorly controlled seizure disorder.

NOTE: A participant with a prior history of seizure could have been considered for enrollment if the Investigator believed the risk of seizure recurrence was low. All cases of prior seizure history were to be discussed with the A5359 protocol leadership team (actg.leada5359@fstrf.org) prior to enrollment.

Advanced liver disease (as defined by any of the following: presence of ascites, encephalopathy, coagulopathy, hypoalbuminemia, esophageal or gastric varices, or persistent jaundice), known biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones) OR history of liver cirrhosis.

Chronic Hepatitis C (HCV) with planned or anticipated use of anti-HCV therapy prior to the completion of Step 2.

History of or current active hepatitis B (HBV) infection defined as a positive HBV surface antigen test or any detectable HBV DNA in participants with isolated HBcAb and HBV DNA as follows:

Participants positive for HBsAg were excluded.

Participants negative for anti-HBs but positive for anti-HBc (negative HBsAg status) and any detectable HBV DNA were excluded.

NOTE: Participants positive for anti-HBc (negative HBsAg status) and positive for anti-HBs (past and/or current evidence) were immune to HBV and were not excluded. If prior documentation of immunity was available, repeat testing at screening was not required.

Current or anticipated need for chronic anti-coagulation therapy.

Unwilling to receive injections, or unable to receive gluteal injections.

Tattoo or other condition over the gluteus region, which could have interfered with the interpretation of injection site reaction.

Previous use of CAB.

Any acute or serious illness, within 7 days prior to entry, requiring systemic treatment and/or hospitalization that could have rendered the participant unable to receive study medication, in the opinion of the site investigator.

QTc greater than 450 ms using either Bazett or Fridericia method within 60 days prior to study entry: Whichever method was used at screening had to be used throughout the study period.

Any serious medical or psychiatric condition, which could have rendered the participant unable to receive study medication in the opinion of the site investigator.

Known allergy/sensitivity or any hypersensitivity to components of study drug(s) or their formulation.

Requirement for any medication that was prohibited with a study medication (refer to protocol-specific web page [PSWP]).

Step 2 Inclusion Criteria

Meeting virologic suppression criteria at or after Step 1, week 4, defined as:

1. HIV-1 RNA ≤200 copies/mL OR
2. HIV-1 RNA of 201-399 copies/mL followed by HIV-1 RNA ≤200 copies/mL by Step 1, week 24.

NOTE: The HIV-1 RNA viral load that was used to determine eligibility for randomization had to have been collected within 4 weeks (28 days) of the Step 2 randomization visit.

Step 2 Exclusion Criteria

Permanent discontinuation of study treatment for any reason during Step 1.

Participants who never started study treatment in Step 1 (see protocol for more information).

Step 3 Inclusion Criteria, Participants Registering from Step 1

Virologic suppression at or after Step 1, week 4, defined as:

1. HIV-1 RNA ≤200 copies/mL OR
2. HIV-1 RNA of 201-399 copies/mL followed by HIV-1 RNA ≤200 copies/mL by Step 1, week 24.

NOTE: The HIV-1 RNA viral load that was used to determine eligibility for Step 3 had to have been collected within 4 weeks (28 days) of the Step 3 registration visit.

Willingness to begin to receive LA ART.

Step 3 Exclusion Criteria, Participants Registering from Step 1

Permanent discontinuation of study treatment for any reason during Step 1.

Participants who never started study treatment in Step 1 (see protocol for more information).

Currently pregnant, planning to become pregnant during the study period, or currently breastfeeding.

Step 3 Inclusion Criteria, Participants Registering from Step 2

Willingness to continue LA ART (for those in Step 2 Arm A) or begin LA ART (for those in Step 2 Arm B).

Step 2 Arm B participants: HIV-1 RNA ≤200 copies/mL at the most recent Step 2 visit OR Confirmation of Virologic Failure visit.

NOTE: The HIV-1 RNA viral load that was used to determine eligibility for Step 3 had to have been collected within 4 weeks (28 days) of the Step 3 registration visit.

Step 3 Exclusion Criteria, Participants Registering from Step 2

Permanent discontinuation of study treatment (LA ART for Arm A and oral ART for Arm B) for any reason during Step 2.

Confirmed Virologic Failure during Step 2.

Step 2 Arm B Participants: Currently pregnant, planning to become pregnant during the study period, or currently breastfeeding.

NOTE: Step 2 Arm A participants who became pregnant and were permitted to continue on LA-ART could continue on that regimen in Step 3.

Step 4 Inclusion Criteria

Any participant who had received at least one dose of CAB-LA or RPV-LA AND did not have access to available LA ART through their provider, OR did not wish to continue LA ART.

Step 4 Exclusion Criteria

There were no exclusion criteria for Step 4.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 456 (Actual)
Dates: Start 2019-03-28 (Actual); Primary Completion 2024-02-12 (Actual); Study Completion 2026-08-30 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Aadia Rana, M.D., Study Chair — Alabama CTU
Locations (33):
- United States (32):
  - Alabama CRS, Birmingham, Alabama
  - University of Southern California CRS, Los Angeles, California
  - UCLA CARE Center CRS, Los Angeles, California
  - UCSD Antiviral Research Center CRS, San Diego, California
  - Ucsf Hiv/Aids Crs, San Francisco, California
  - Harbor-UCLA CRS, Torrance, California
  - University of Colorado Hospital CRS, Aurora, Colorado
  - Univ. of Florida Jacksonville NICHD CRS, Jacksonville, Florida
  - The Ponce de Leon Center CRS, Atlanta, Georgia
  - Northwestern University CRS, Chicago, Illinois
  - Rush University CRS, Chicago, Illinois
  - Johns Hopkins University CRS, Baltimore, Maryland
  - Massachusetts General Hospital CRS (MGH CRS), Boston, Massachusetts
  - Brigham and Women's Hospital Therapeutics Clinical Research Site (BWH TCRS) CRS, Boston, Massachusetts
  - Washington University Therapeutics (WT) CRS, St Louis, Missouri
  - New Jersey Medical School Clinical Research Center CRS, Newark, New Jersey
  - Weill Cornell Chelsea CRS, New York, New York
  - Columbia P&S CRS, New York, New York
  - Weill Cornell Uptown CRS, New York, New York
  - SUNY Stony Brook NICHD CRS, Stony Brook, New York
  - Jacobi Med. Ctr. Bronx NICHD CRS, The Bronx, New York
  - Chapel Hill CRS, Chapel Hill, North Carolina
  - Greensboro CRS, Greensboro, North Carolina
  - Cincinnati Clinical Research Site, Cincinnati, Ohio
  - Case Clinical Research Site, Cleveland, Ohio
  - Ohio State University CRS, Columbus, Ohio
  - Penn Therapeutics, CRS, Philadelphia, Pennsylvania
  - University of Pittsburgh CRS, Pittsburgh, Pennsylvania
  - The Miriam Hospital Clinical Research Site (TMH CRS) CRS, Providence, Rhode Island
  - Vanderbilt Therapeutics (VT) CRS, Nashville, Tennessee
  - Houston AIDS Research Team CRS, Houston, Texas
  - University of Washington AIDS CRS, Seattle, Washington
- Puerto Rico AIDS Clinical Trials Unit CRS, San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie results in the publication, after deidentification.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 3 months following publication and available throughout period of funding of the AIDS Clinical Trials Group by NIH.
Access Criteria: * With whom?
    * Researchers who provide a methodologically sound proposal for use of the data that is approved by the AIDS Clinical Trials Group.
  * For what types of analyses?
    * To achieve aims in the proposal approved by the AIDS Clinical Trials Group.
  * By what mechanism will data be made available?
    * Researchers may submit a request for access to data using the AIDS Clinical Trials Group "Data Request" form at: https://submit.mis.s-3.net/. Researchers of approved proposals will need to sign an AIDS Clinical Trials Group Data Use Agreement before receiving the data.

REFERENCES:
- [Derived] Okesanya OJ, Ayeni RA, Amadin P, Ngwoke I, Amisu BO, Ukoaka BM, Ahmed MM, Oso TA, Musa SS, Lucero-Prisno DE. Advances in HIV Treatment and Vaccine Development: Emerging Therapies and Breakthrough Strategies for Long-Term Control. AIDS Res Treat. 2025 Jul 4;2025:6829446. doi: 10.1155/arat/6829446. eCollection 2025. PMID 40655875
- [Derived] Pluznik JA, Nijhawan AE, Spaulding AC. Does Anything Work? Improving HIV Care Engagement for Individuals Transitioning out of Correctional Settings. J Acquir Immune Defic Syndr. 2021 Mar 1;86(3):286-287. doi: 10.1097/QAI.0000000000002599. No abstract available. PMID 33560746
- See also: The Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE Grading Table), Version 1.0, December 2004 (Clarification, August 2009). — https://rsc.niaid.nih.gov/sites/default/files/daidsgradingcorrectedv21.pdf
- See also: Manual for Expedited Reporting of Adverse Events to DAIDS (DAIDS EAE Manual), Version 2.0, January 2010 — https://rsc.niaid.nih.gov/sites/default/files/manual-exped-aes-v2_0.pdf
- See also: FDA Snapshot algorithm — https://www.fda.gov/files/drugs/published/Human-Immunodeficiency-Virus-1-Infection--Developing-Antiretroviral-Drugs-for-Treatment.pdf
- See also: IAS October/November 2022 Update of the Drug Resistance Mutations in HIV-1 — https://www.iasusa.org/wp-content/uploads/2022/10/30-4-559.pdf
- See also: Alcohol Use Disorders Identification Test — https://www.hepatitis.va.gov/alcohol/treatment/audit-c.asp

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 33 Clinical Research Sites (CRSs) in the United States between March 28, 2019 and February 12, 2024. A total of 456 participants enrolled to study. After completing Step 1, 308 participants were randomized to Step 2. Enrollment to Step 3 and Step 4 will be updated upon study completion.
Pre-assignment Details: Step 1 eligibility violations were identified in three participants. One participant was found to have missed the screening confirmatory HBV DNA test. Two participants were found to have past exclusionary mutations after enrolled to Step 2. All three participants were excluded from all analyses. 453 eligible participants were enrolled to Step 1. 306 eligible participants were randomized to Step 2 after completing Step 1.
Groups:
- Step 2 Arm A: LA-ART: In Step 2, participants received oral RPV once daily and oral CAB once daily for 4 weeks (optional), followed by a RPV-LA loading dose and a CAB-LA loading dose, followed in 4 weeks by an RPV-LA maintenance dose and a CAB-LA maintenance dose every 4 weeks for 44 weeks.
Period: Step 1
Arm/Group | Step 1 SOC | Step 2 Arm A: LA-ART | Step 2 Arm B: SOC
Started | 453 | 0 | 0
Completed | 360 | 0 | 0
Not Completed | 93 | 0 | 0
Not completed — Death | 1 | 0 | 0
Not completed — Lost to Follow-up | 31 | 0 | 0
Not completed — Pregnancy | 1 | 0 | 0
Not completed — Protocol Violation | 8 | 0 | 0
Not completed — Withdrawal by Subject | 13 | 0 | 0
Not completed — Other reasons | 12 | 0 | 0
Not completed — On Step 1 as of February 12, 2024 | 27 | 0 | 0
Period: Step 2
Arm/Group | Step 1 SOC | Step 2 Arm A: LA-ART | Step 2 Arm B: SOC
Started | 0 | 152 | 154
Completed | 0 | 76 | 74
Not Completed | 0 | 76 | 80
Not completed — Lost to Follow-up | 0 | 8 | 15
Not completed — Withdrawal by Subject | 0 | 6 | 6
Not completed — Death | 0 | 2 | 0
Not completed — Incarceration | 0 | 2 | 0
Not completed — Non-Compliance With Study Requirements | 0 | 1 | 1
Not completed — Confounding Medical Condition | 0 | 0 | 1
Not completed — Out Of State With No Plan To Return | 0 | 1 | 0
Not completed — Switched To Injectables | 0 | 0 | 1
Not completed — On Step 2 as of February 12, 2024 | 0 | 56 | 56

BASELINE CHARACTERISTICS:
Population: Step 1 baseline analysis population was defined as all eligible participants who registered to Step 1. Step 2 baseline analysis population was defined as all eligible participants who were randomized to the treatment arms, regardless of status on randomized treatment.
Groups:
- Step 2 Arm B: SOC: In Step 2, participants received SOC oral ART regimen for 52 weeks.
- Total: Total of all reporting groups
Arm/Group | Step 1 SOC | Step 2 Arm A: LA-ART | Step 2 Arm B: SOC | Total
Number analyzed (Participants) | 453 | 152 | 154 | 759
Age, Continuous [Median (Inter-Quartile Range); unit: years] — Population: Step 1 baseline measurement included 453 participants who were enrolled in the study. Step 2 baseline measurement included 306 participants who were randomized to Step 2.
  years
    Step 1: number analyzed (Participants) | 453 | 0 | 0 | 453
    Step 1 | 40 [32 to 51] |  |  | 40 [32 to 51]
    Step 2: number analyzed (Participants) | 0 | 152 | 154 | 306
    Step 2 |  | 41 [32 to 53] | 42 [33 to 52] | 42 [32 to 52]
Age, Customized [Count of Participants; unit: Participants] — Population: Step 1 baseline measurement included 453 participants who were enrolled in the study. Step 2 baseline measurement included 306 participants who were randomized to Step 2.
  Participants
    Step 1: number analyzed (Participants) | 453 | 0 | 0 | 453
    Step 1: 18-24 | 29 |  |  | 29
    Step 1: 25-30 | 64 |  |  | 64
    Step 1: 31-40 | 142 |  |  | 142
    Step 1: 41-50 | 102 |  |  | 102
    Step 1: 51+ | 116 |  |  | 116
    Step 2: number analyzed (Participants) | 0 | 152 | 154 | 306
    Step 2: 18-24 |  | 8 | 7 | 15
    Step 2: 25-30 |  | 21 | 20 | 41
    Step 2: 31-40 |  | 46 | 40 | 86
    Step 2: 41-50 |  | 27 | 45 | 72
    Step 2: 51+ |  | 50 | 42 | 92
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Step 1 baseline measurement included 453 participants who were enrolled in the study. Step 2 baseline measurement included 306 participants who were randomized to Step 2.
  Participants
    Step 1: number analyzed (Participants) | 453 | 0 | 0 | 453
    Step 1: Female | 133 |  |  | 133
    Step 1: Male | 320 |  |  | 320
    Step 2: number analyzed (Participants) | 0 | 152 | 154 | 306
    Step 2: Female |  | 43 | 41 | 84
    Step 2: Male |  | 109 | 113 | 222
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Step 1 baseline measurement included 453 participants who were enrolled in the study. Step 2 baseline measurement included 306 participants who were randomized to Step 2.
  Participants
    Step 1: number analyzed (Participants) | 453 | 0 | 0 | 453
    Step 1: Hispanic or Latino | 79 |  |  | 79
    Step 1: Not Hispanic or Latino | 369 |  |  | 369
    Step 1: Unknown or Not Reported | 5 |  |  | 5
    Step 2: number analyzed (Participants) | 0 | 152 | 154 | 306
    Step 2: Hispanic or Latino |  | 29 | 26 | 55
    Step 2: Not Hispanic or Latino |  | 121 | 125 | 246
    Step 2: Unknown or Not Reported |  | 2 | 3 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Step 1 baseline measurement included 453 participants who were enrolled in the study. Step 2 baseline measurement included 306 participants who were randomized to Step 2.
  Participants
    Step 1: number analyzed (Participants) | 453 | 0 | 0 | 453
    Step 1: American Indian or Alaska Native | 0 |  |  | 0
    Step 1: Asian | 3 |  |  | 3
    Step 1: Native Hawaiian or Other Pacific Islander | 0 |  |  | 0
    Step 1: Black or African American | 286 |  |  | 286
    Step 1: White | 125 |  |  | 125
    Step 1: More than one race | 11 | 0 |  | 11
    Step 1: Unknown or Not Reported | 28 | 0 |  | 28
    Step 2: number analyzed (Participants) | 0 | 152 | 154 | 306
    Step 2: American Indian or Alaska Native |  | 0 | 0 | 0
    Step 2: Asian |  | 1 | 1 | 2
    Step 2: Native Hawaiian or Other Pacific Islander |  | 0 | 0 | 0
    Step 2: Black or African American |  | 94 | 103 | 197
    Step 2: White |  | 44 | 36 | 80
    Step 2: More than one race |  | 4 | 2 | 6
    Step 2: Unknown or Not Reported |  | 9 | 12 | 21
History of IV drug use [Count of Participants; unit: Participants] — Population: Step 1 baseline measurement included 453 participants who were enrolled in the study. Step 2 baseline measurement included 306 participants who were randomized to Step 2.
  Participants
    Step 1: number analyzed (Participants) | 453 | 0 | 0 | 453
    Step 1: Currently | 20 |  |  | 20
    Step 1: Previously | 43 |  |  | 43
    Step 1: Never | 390 |  |  | 390
    Step 2: number analyzed (Participants) | 0 | 152 | 154 | 306
    Step 2: Currently |  | 8 | 4 | 12
    Step 2: Previously |  | 15 | 12 | 27
    Step 2: Never |  | 129 | 138 | 267
BMI, continuous [Median (Inter-Quartile Range); unit: kg/m²] — Population: Step 1 baseline measurement included 453 participants who were enrolled in the study. Step 2 baseline measurement included 306 participants who were randomized to Step 2.
  kg/m²
    Step 1: number analyzed (Participants) | 453 | 0 | 0 | 453
    Step 1 | 26 [22 to 30] |  |  | 26 [22 to 30]
    Step 2: number analyzed (Participants) | 0 | 152 | 154 | 306
    Step 2 |  | 27 [23 to 31] | 26 [23 to 31] | 26 [23 to 31]
Time since HIV diagnosis [Median (Inter-Quartile Range); unit: years] — Population: Step 1 baseline measurement included 453 participants who were enrolled in the study. Step 2 baseline measurement included 306 participants who were randomized to Step 2.
  years
    Step 1: number analyzed (Participants) | 453 | 0 | 0 | 453
    Step 1 | 13 [7 to 21] |  |  | 13 [7 to 21]
    Step 2: number analyzed (Participants) | 0 | 152 | 154 | 306
    Step 2 |  | 13 [7 to 22] | 12 [7 to 19] | 13 [7 to 20]
Non-Adherence information [Count of Participants; unit: Participants] — Population: Step 1 baseline measurement included 453 participants who were enrolled in the study. Step 2 baseline measurement included 306 participants who were randomized to Step 2.
  Participants
    Step 1: number analyzed (Participants) | 453 | 0 | 0 | 453
    Step 1: Lost to follow-up | 93 |  |  | 93
    Step 1: Poor virologic response | 294 |  |  | 294
    Step 1: Poor virologic response and lost to follow-up | 66 |  |  | 66
    Step 2: number analyzed (Participants) | 0 | 152 | 154 | 306
    Step 2: Lost to follow-up |  | 33 | 37 | 70
    Step 2: Poor virologic response |  | 99 | 95 | 194
    Step 2: Poor virologic response and lost to follow-up |  | 20 | 22 | 42
HIV-1 RNA levels, categorical [Count of Participants; unit: Participants] — Population: Step 1 baseline measurement included 453 participants who were enrolled in the study. Step 2 baseline measurement included 306 participants who were randomized to Step 2.
  Participants
    Step 1: number analyzed (Participants) | 453 | 0 | 0 | 453
    Step 1: <50 | 85 |  |  | 85
    Step 1: 50-200 | 69 |  |  | 69
    Step 1: 201-399 | 16 |  |  | 16
    Step 1: 400-1,000 | 28 |  |  | 28
    Step 1: 1,001-5,000 | 48 |  |  | 48
    Step 1: 5,001-10,000 | 22 |  |  | 22
    Step 1: >10,000 | 123 |  |  | 123
    Step 1: Not done | 58 |  |  | 58
    Step 1: Missing | 4 |  |  | 4
    Step 2: number analyzed (Participants) | 0 | 152 | 154 | 306
    Step 2: <50 |  | 108 | 123 | 231
    Step 2: 50-200 |  | 18 | 19 | 37
    Step 2: 201-399 |  | 5 | 3 | 8
    Step 2: 400-1,000 |  | 4 | 3 | 7
    Step 2: 1,001-5,000 |  | 6 | 2 | 8
    Step 2: 5,001-10,000 |  | 1 | 1 | 2
    Step 2: >10,000 |  | 8 | 1 | 9
    Step 2: Not done |  | 2 | 1 | 3
    Step 2: Missing |  | 0 | 1 | 1
Step 1 HIV-1 RNA, continuous [Median (Inter-Quartile Range); unit: log10 copies/mL] — Population: Step 1 baseline measurement included 453 participants who were enrolled in the study.
  log10 copies/mL
    number analyzed (Participants) | 453 | 0 | 0 | 453
    (all) | 3.45 [1.91 to 4.57] |  |  | 3.45 [1.91 to 4.57]
Step 2 HIV-1 RNA levels, categorical [Count of Participants; unit: Participants] — Population: Step 2 baseline measurement included 306 participants who were randomized to Step 2.
  Participants
    number analyzed (Participants) | 0 | 152 | 154 | 306
    ≤200 |  | 126 | 142 | 268
    >200 |  | 24 | 10 | 34
    Not done |  | 2 | 1 | 3
    Missing |  | 0 | 1 | 1
CD4, continuous [Median (Inter-Quartile Range); unit: cells/mm^3] — Population: Step 1 baseline measurement included 453 participants who were enrolled in the study. Step 2 baseline measurement included 306 participants who were randomized to Step 2.
  cells/mm^3
    Step 1: number analyzed (Participants) | 453 | 0 | 0 | 453
    Step 1 | 273 [119 to 511] |  |  | 273 [119 to 511]
    Step 2: number analyzed (Participants) | 0 | 152 | 154 | 306
    Step 2 |  | 417 [198 to 703] | 379 [202 to 611] | 389 [199 to 638]
CD8, continuous [Median (Inter-Quartile Range); unit: cells/mm^3] — Population: Step 1 baseline measurement included 453 participants who were enrolled in the study. Step 2 baseline measurement included 306 participants who were randomized to Step 2.
  cells/mm^3
    Step 1: number analyzed (Participants) | 453 | 0 | 0 | 453
    Step 1 | 843 [586 to 1225] |  |  | 843 [586 to 1225]
    Step 2: number analyzed (Participants) | 0 | 152 | 154 | 306
    Step 2 |  | 846 [630 to 1140] | 866 [615 to 1254] | 861 [616 to 1179]
Education Level [Count of Participants; unit: Participants] — Population: Step 1 baseline measurement included 453 participants who were enrolled in the study. Step 2 baseline measurement included 306 participants who were randomized to Step 2.
  Participants
    Step 1: number analyzed (Participants) | 453 | 0 | 0 | 453
    Step 1: 11th grade or less | 89 |  |  | 89
    Step 1: High school graduate or GED | 141 |  |  | 141
    Step 1: Some college/AA degree/Technical school training | 162 |  |  | 162
    Step 1: College graduate (BA or BS) | 40 |  |  | 40
    Step 1: Master's degree | 6 |  |  | 6
    Step 1: Doctorate/medical degree/law degree | 6 |  |  | 6
    Step 1: Missing | 9 |  |  | 9
    Step 2: number analyzed (Participants) | 0 | 152 | 154 | 306
    Step 2: 11th grade or less |  | 32 | 27 | 59
    Step 2: High school graduate or GED |  | 47 | 48 | 95
    Step 2: Some college/AA degree/Technical school training |  | 54 | 54 | 108
    Step 2: College graduate (BA or BS) |  | 11 | 13 | 24
    Step 2: Master's degree |  | 1 | 5 | 6
    Step 2: Doctorate/medical degree/law degree |  | 2 | 3 | 5
    Step 2: Missing |  | 5 | 4 | 9
Employment or School [Count of Participants; unit: Participants] — Population: Step 1 baseline measurement included 453 participants who were enrolled in the study. Step 2 baseline measurement included 306 participants who were randomized to Step 2.
  Participants
    Step 1: number analyzed (Participants) | 453 | 0 | 0 | 453
    Step 1: Part-time employment | 61 |  |  | 61
    Step 1: Full-time employment | 117 |  |  | 117
    Step 1: Part-time student | 3 |  |  | 3
    Step 1: Full-time student | 13 |  |  | 13
    Step 1: On disability | 96 |  |  | 96
    Step 1: Pension/Retired | 11 |  |  | 11
    Step 1: OTHER | 147 |  |  | 147
    Step 1: Missing | 5 |  |  | 5
    Step 2: number analyzed (Participants) | 0 | 152 | 154 | 306
    Step 2: Part-time employment |  | 23 | 17 | 40
    Step 2: Full-time employment |  | 45 | 49 | 94
    Step 2: Part-time student |  | 1 | 1 | 2
    Step 2: Full-time student |  | 3 | 2 | 5
    Step 2: On disability |  | 28 | 35 | 63
    Step 2: Pension/Retired |  | 6 | 3 | 9
    Step 2: OTHER |  | 43 | 44 | 87
    Step 2: Missing |  | 3 | 3 | 6
Average Yearly Household Income [Count of Participants; unit: Participants] — Population: Step 1 baseline measurement included 453 participants who were enrolled in the study. Step 2 baseline measurement included 306 participants who were randomized to Step 2.
  Participants
    Step 1: number analyzed (Participants) | 453 | 0 | 0 | 453
    Step 1: Less than $5000 per year | 128 |  |  | 128
    Step 1: $5000 - 9999 | 59 |  |  | 59
    Step 1: $10000 - 19999 | 99 |  |  | 99
    Step 1: $20000 - 29999 | 54 |  |  | 54
    Step 1: $30000 - 39999 | 45 |  |  | 45
    Step 1: $40000 - 49999 | 28 |  |  | 28
    Step 1: $50000 or more per year | 26 |  |  | 26
    Step 1: Missing | 14 |  |  | 14
    Step 2: number analyzed (Participants) | 0 | 152 | 154 | 306
    Step 2: Less than $5000 per year |  | 42 | 47 | 89
    Step 2: $5000 - 9999 |  | 24 | 22 | 46
    Step 2: $10000 - 19999 |  | 32 | 31 | 63
    Step 2: $20000 - 29999 |  | 17 | 16 | 33
    Step 2: $30000 - 39999 |  | 18 | 15 | 33
    Step 2: $40000 - 49999 |  | 8 | 4 | 12
    Step 2: $50000 or more per year |  | 8 | 16 | 24
    Step 2: Missing |  | 3 | 3 | 6
How to Pay Healthcare [Count of Participants; unit: Participants] — Population: Step 1 baseline measurement included 453 participants who were enrolled in the study. Step 2 baseline measurement included 306 participants who were randomized to Step 2.
  Participants
    Step 1: number analyzed (Participants) | 453 | 0 | 0 | 453
    Step 1: Government Funding | 350 |  |  | 350
    Step 1: Government Funding, Private Insurance | 15 |  |  | 15
    Step 1: Government Funding, Private Insurance, Self Pay/Out of Pocket | 3 |  |  | 3
    Step 1: Government Funding, Self Pay/Out of Pocket | 20 |  |  | 20
    Step 1: Private Insurance | 30 |  |  | 30
    Step 1: Private Insurance, Self Pay/Out of Pocket | 3 |  |  | 3
    Step 1: Self Pay/Out of Pocket | 12 |  |  | 12
    Step 1: Missing | 20 |  |  | 20
    Step 2: number analyzed (Participants) | 0 | 152 | 154 | 306
    Step 2: Government Funding |  | 117 | 112 | 229
    Step 2: Government Funding, Private Insurance |  | 4 | 10 | 14
    Step 2: Government Funding, Private Insurance, Self Pay/Out of Pocket |  | 2 | 2 | 4
    Step 2: Government Funding, Self Pay/Out of Pocket |  | 7 | 4 | 11
    Step 2: Private Insurance |  | 8 | 12 | 20
    Step 2: Private Insurance, Self Pay/Out of Pocket |  | 0 | 2 | 2
    Step 2: Self Pay/Out of Pocket |  | 6 | 5 | 11
    Step 2: Missing |  | 8 | 7 | 15
Provide Support to Friend/Family Member [Count of Participants; unit: Participants] — Population: Step 1 baseline measurement included 453 participants who were enrolled in the study. Step 2 baseline measurement included 306 participants who were randomized to Step 2.
  Participants
    Step 1: number analyzed (Participants) | 453 | 0 | 0 | 453
    Step 1: Yes | 116 |  |  | 116
    Step 1: No | 332 |  |  | 332
    Step 1: Missing | 5 |  |  | 5
    Step 2: number analyzed (Participants) | 0 | 152 | 154 | 306
    Step 2: Yes |  | 41 | 40 | 81
    Step 2: No |  | 109 | 112 | 221
    Step 2: Missing |  | 2 | 2 | 4
Living Situation [Count of Participants; unit: Participants] — Population: Step 1 baseline measurement included 453 participants who were enrolled in the study. Step 2 baseline measurement included 306 participants who were randomized to Step 2.
  Participants
    Step 1: number analyzed (Participants) | 453 | 0 | 0 | 453
    Step 1: In Own House/Apartment | 270 |  |  | 270
    Step 1: At Parents House | 64 |  |  | 64
    Step 1: Someone Else House/Apartment | 57 |  |  | 57
    Step 1: Rooming Boarding Or Halfway House | 17 |  |  | 17
    Step 1: Shelter/Welfare Hotel | 15 |  |  | 15
    Step 1: On The Street(S) | 9 |  |  | 9
    Step 1: Residential Drug/Alcohol Treatment Facility | 1 |  |  | 1
    Step 1: Other | 11 |  |  | 11
    Step 1: Missing | 9 |  |  | 9
    Step 2: number analyzed (Participants) | 0 | 152 | 154 | 306
    Step 2: In Own House/Apartment |  | 101 | 99 | 200
    Step 2: At Parents House |  | 15 | 21 | 36
    Step 2: Someone Else House/Apartment |  | 25 | 16 | 41
    Step 2: Rooming Boarding Or Halfway House |  | 1 | 5 | 6
    Step 2: Shelter/Welfare Hotel |  | 3 | 6 | 9
    Step 2: On The Street(S) |  | 1 | 3 | 4
    Step 2: Residential Drug/Alcohol Treatment Facility |  | 2 | 0 | 2
    Step 2: Other |  | 2 | 2 | 4
    Step 2: Missing |  | 2 | 2 | 4
Treated for Depression or Mental Health [Count of Participants; unit: Participants] — Population: Step 1 baseline measurement included 453 participants who were enrolled in the study. Step 2 baseline measurement included 306 participants who were randomized to Step 2.
  Participants
    Step 1: number analyzed (Participants) | 453 | 0 | 0 | 453
    Step 1: Yes | 124 |  |  | 124
    Step 1: No | 323 |  |  | 323
    Step 1: Missing | 6 |  |  | 6
    Step 2: number analyzed (Participants) | 0 | 152 | 154 | 306
    Step 2: Yes |  | 41 | 36 | 77
    Step 2: No |  | 109 | 116 | 225
    Step 2: Missing |  | 2 | 2 | 4
Smoke Status [Count of Participants; unit: Participants] — Population: Step 1 baseline measurement included 453 participants who were enrolled in the study. Step 2 baseline measurement included 306 participants who were randomized to Step 2.
  Participants
    Step 1: number analyzed (Participants) | 453 | 0 | 0 | 453
    Step 1: NEVER | 143 |  |  | 143
    Step 1: FORMER | 89 |  |  | 89
    Step 1: CUREENT | 220 |  |  | 220
    Step 1: Missing | 1 |  |  | 1
    Step 2: number analyzed (Participants) | 0 | 152 | 154 | 306
    Step 2: NEVER |  | 47 | 57 | 104
    Step 2: FORMER |  | 27 | 34 | 61
    Step 2: CUREENT |  | 78 | 63 | 141
    Step 2: Missing |  | 0 | 0 | 0
Participant Health Questionnaire (PHQ-9) total score [0-27] [Count of Participants; unit: Participants] — The Participant Health Questionnaire consists of 9 items scored as follows: 0 = Not at all, 1 = Several days, 2 = More than half the days, 3 = Nearly every day. Population: Step 1 baseline measurement included 453 participants who were enrolled in the study. Step 2 baseline measurement included 306 participants who were randomized to Step 2.
  Participants
    Step 1: number analyzed (Participants) | 453 | 0 | 0 | 453
    Step 1: No Depression [0-4] | 228 |  |  | 228
    Step 1: Mild Depression [5-9] | 106 |  |  | 106
    Step 1: Moderate Depression [10-14] | 56 |  |  | 56
    Step 1: Severe Depression [15-27] | 60 |  |  | 60
    Step 1: Missing | 3 |  |  | 3
    Step 2: number analyzed (Participants) | 0 | 152 | 154 | 306
    Step 2: No Depression [0-4] |  | 85 | 89 | 174
    Step 2: Mild Depression [5-9] |  | 29 | 35 | 64
    Step 2: Moderate Depression [10-14] |  | 24 | 20 | 44
    Step 2: Severe Depression [15-27] |  | 14 | 10 | 24
    Step 2: Missing |  | 0 | 0 | 0
General Anxiety Disorder (GAD-7) [Count of Participants; unit: Participants] — Population: Step 1 baseline measurement included 453 participants who were enrolled in the study. Step 2 baseline measurement included 306 participants who were randomized to Step 2.
  Participants
    Step 1: number analyzed (Participants) | 453 | 0 | 0 | 453
    Step 1: No Anxiety [<5] | 228 |  |  | 228
    Step 1: Mild [5-<10] | 106 |  |  | 106
    Step 1: Moderate [10-<15] | 56 |  |  | 56
    Step 1: Severe Anxiety [15+] | 60 |  |  | 60
    Step 1: Missing | 3 |  |  | 3
    Step 2: number analyzed (Participants) | 0 | 152 | 154 | 306
    Step 2: No Anxiety [<5] |  | 84 | 76 | 160
    Step 2: Mild [5-<10] |  | 38 | 46 | 84
    Step 2: Moderate [10-<15] |  | 18 | 22 | 40
    Step 2: Severe Anxiety [15+] |  | 12 | 10 | 22
    Step 2: Missing |  | 0 | 0 | 0
Suicide Severity Rating [Count of Participants; unit: Participants] — Population: Step 1 baseline measurement included 453 participants who were enrolled in the study. Step 2 baseline measurement included 306 participants who were randomized to Step 2.
  Participants
    Step 1: number analyzed (Participants) | 453 | 0 | 0 | 453
    Step 1: No Risk | 358 |  |  | 358
    Step 1: Low Risk | 31 |  |  | 31
    Step 1: Moderate Risk | 45 |  |  | 45
    Step 1: High Risk | 10 |  |  | 10
    Step 1: Missing | 9 |  |  | 9
    Step 2: number analyzed (Participants) | 0 | 152 | 154 | 306
    Step 2: No Risk |  | 125 | 129 | 254
    Step 2: Low Risk |  | 12 | 7 | 19
    Step 2: Moderate Risk |  | 14 | 13 | 27
    Step 2: High Risk |  | 1 | 1 | 2
    Step 2: Missing |  | 0 | 4 | 4
Drug Dependency [Count of Participants; unit: Participants] — Drug Dependency is defined as: No Drug Problems [<6 for male and <2 for female]; Drug-Use-Related problems [between [6, 25) for male and [2, 25) for female]), Drug Dependency [>=25 regardless of sex] by Drug Use Disorders Identification Test result. Population: Step 1 baseline measurement included 453 participants who were enrolled in the study. Step 2 baseline measurement included 306 participants who were randomized to Step 2.
  Participants
    Step 1: number analyzed (Participants) | 453 | 0 | 0 | 453
    Step 1: No Drug Problems | 224 |  |  | 224
    Step 1: Drug-Use-Related Problems | 205 |  |  | 205
    Step 1: Drug Dependency | 23 |  |  | 23
    Step 1: Missing | 1 |  |  | 1
    Step 2: number analyzed (Participants) | 0 | 152 | 154 | 306
    Step 2: No Drug Problems |  | 76 | 83 | 159
    Step 2: Drug-Use-Related Problems |  | 69 | 64 | 133
    Step 2: Drug Dependency |  | 7 | 7 | 14
    Step 2: Missing |  | 0 | 0 | 0
AUDIT-C Alcohol Consumption Score [Median (Inter-Quartile Range); unit: score] — 3 alcohol consumption questions:
  1. How often did you have a drink containing alcohol in the past year?
  2. On days in the past year when you drank alcohol how many drinks did you typically drink?
  3. How often did you have 6 or more (for men) or 4 or more (for women and everyone 65 and older) drinks on an occasion in the past year?
  The minimum score (for non-drinkers) is 0 and the maximum possible score is 12. Population: Step 1 baseline measurement included 453 participants who were enrolled in the study. Step 2 baseline measurement included 306 participants who were randomized to Step 2.
  score
    Step 1: number analyzed (Participants) | 453 | 0 | 0 | 453
    Step 1 | 2 [1 to 4] |  |  | 2 [1 to 4]
    Step 2: number analyzed (Participants) | 0 | 152 | 154 | 306
    Step 2 |  | 2 [0 to 3] | 2 [0 to 4] | 2 [0 to 4]

OUTCOME MEASURES:

1. Primary Outcome: Cumulative Probability of Regimen Failure in Step 2 at Any Time Post Randomization and Week 48 Visit
Description: Regimen failure was defined as the occurrence of the earlier of the following two events
  * virologic failure (defined as two consecutive HIV-1 RNA >200 copies/mL after Step 2 randomization
  * Permanent discontinuation of randomized study treatment prior to or at Week 48 visit
  Cumulative probability was calculated by Kaplan-Meier method.
Time Frame: From Step 2 randomization to Step 2, Week 48 visit (up to 50 weeks)
Population: Intention-to-Treat (ITT) Population was defined as all eligible participants who were randomized to the treatment arms, regardless of status on randomized treatment. Participants were assessed according to their randomized treatment, regardless of the treatment they received.
Measure: Number; unit: cumulative percent probability of event
Arm/Group | Step 2 Arm A: LA ART | Step 2 Arm B: SOC
Number analyzed (Participants) | 152 | 154
cumulative percent probability of event | 22.8 | 41.2
Statistical Analysis 1: Comparison: Step 2 Arm A: LA ART vs Step 2 Arm B: SOC; Treatment comparison was conducted by cumulative probability of regimen failure in Step 2 up to Step 2 Week 48 visit by treatment arm. The treatment difference was assessed using the 95% repeated confidence interval adjusted for interim efficacy analyses, i.e., a nominal 98.4% confidence interval; Test type: Superiority — The study had approximately 80% power to show superiority of the LA ART compared to daily SOC with respect to the Step 2, week 48, cumulative probability of regimen failure; Cumulative probability difference = -18.4, 98.4% CI 2-sided [-32.4 to -4.3] — Treatment difference was calculated as LA-ART minus SOC. 98.4% is nominal confidence interval

2. Secondary Outcome: Cumulative Probability of Virologic Failure in Step 2 at Any Time Post Randomization to Week 48 Visit
Description: Virologic failure was defined as two consecutive HIV-1 RNA >200 copies/mL after Step 2 randomization and up to Step 2 Week 48 visit, regardless of the time between them.
  Cumulative probability was calculated by Kaplan-Meier method.
Time Frame: From Step 2 randomization to Step 2, Week 48 visit (up to 50 weeks)
Population: as for outcome 1
Measure: Number; unit: cumulative percent probability of event
Arm/Group | Step 2 Arm A: LA ART | Step 2 Arm B: SOC
Number analyzed (Participants) | 152 | 154
cumulative percent probability of event | 6.8 | 28.2
Statistical Analysis 1: Comparison: Step 2 Arm A: LA ART vs Step 2 Arm B: SOC; Treatment comparison was conducted by cumulative probability of virologic failure in Step 2 up to Step 2 Week 48 visit by treatment arm. The treatment difference was assessed using the 95% repeated confidence interval adjusted for interim efficacy analyses, i.e., a nominal 98.4% confidence interval; Test type: Superiority — The study had at least 80% power to show superiority of the LA ART compared to daily SOC with respect to the Step 2, week 48, cumulative probability of virologic failure; cumulative probability difference = -21.4, 98.4% CI 2-sided [-33.5 to -9.3] — Treatment difference was calculated as LA-ART minus SOC.98.4% is nominal confidence interval

3. Secondary Outcome: Cumulative Probability of the Treatment-related Failure in Step 2 at Any Time Post Randomization to Week 48 Visit
Description: Treatment-related failure was defined as the occurrence of the earlier of virologic failure or permanent Step 2 treatment discontinuation due to treatment-related adverse events.
  Cumulative probability was calculated by Kaplan-Meier method.
Time Frame: From after Step 2 randomization to Step 2, Week 48 (up to 50 weeks)
Population: as for outcome 1
Measure: Number; unit: cumulative percent probability of event
Arm/Group | Step 2 Arm A: LA ART | Step 2 Arm B: SOC
Number analyzed (Participants) | 152 | 154
cumulative percent probability of event | 8.9 | 28.1
Statistical Analysis 1: Comparison: Step 2 Arm A: LA ART vs Step 2 Arm B: SOC; Treatment comparison was conducted by cumulative probability of treatment-related failure in Step 2 up to Step 2 Week 48 visit by treatment arm. The treatment difference was assessed using the 95% repeated confidence interval adjusted for interim efficacy analyses, i.e., a nominal 98.4% confidence interval; Test type: Superiority; cumulative probability diffeence = -19.2, 98.4% CI 2-sided [-31.6 to -6.9]; Treatment difference was calculated as LA-ART minus SOC.98.4% is nominal confidence interval

4. Secondary Outcome: Number of Participants With Virologic Non-success (>= 50 Copies/ml)
Description: Virologic non-success was defined by the US Food and Drug Administration (FDA) Snapshot algorithm
Time Frame: from Step 2 randomization to Step 2, Week 48 (up to 50 weeks)
Population: The analysis population was restricted to participants randomized at least 50 weeks prior to February 12, 2024.
Measure: Count of Participants; unit: Participants
Arm/Group | Step 2 Arm A: LA ART | Step 2 Arm B: SOC
Number analyzed (Participants) | 94 | 96
Participants
  HIV-1 RNA < 50 copies/ml | 62 | 49
  HIV-1 RNA >= 50 copies/ml | 14 | 33
  Treatment Discontinuation due to AE or Death | 6 | 0
  Treatment Discontinuation due to other reasons with HIV-1 RNA < 50 copies/ml | 10 | 13
  On treatment but missing data | 2 | 1
Statistical Analysis 1: Comparison: Step 2 Arm A: LA ART vs Step 2 Arm B: SOC; Test type: Superiority — The proportions of participants with HIV-1 RNA ≥ 50 copies/ml was compared by Fisher's Exact Test; p < 0.001, Fisher Exact; Mean Difference (Final Values) = -21.8, 95% CI 2-sided [-35.6 to -8.1]; Treatment difference in the proportions of participants with HIV-1 RNA ≥ 50 copies/ml was calculated as LA-ART minus SOC

5. Secondary Outcome: Number of Participants With Virologic Non-success (>= 200 Copies/ml)
Description: Virologic non-success was defined by the US Food and Drug Administration (FDA) Snapshot algorithm
Time Frame: From Step 2 randomization to Step 2, Week 48 (up to 50 weeks)
Population: The analysis population was restricted to participants randomized at least 50 weeks prior to February 12, 2024.
Measure: Count of Participants; unit: Participants
Arm/Group | Step 2 Arm A: LA ART | Step 2 Arm B: SOC
Number analyzed (Participants) | 94 | 96
Participants
  HIV-1 RNA < 200 copies/ml | 69 | 55
  HIV-1 RNA >= 200 copies/ml | 5 | 25
  Treatment Discontinuation due to AE or Death | 6 | 0
  Treatment Discontinuation due to other reasons with HIV-1 RNA < 200 copies/ml | 12 | 15
  On treatment but missing data | 2 | 1
Statistical Analysis 1: Comparison: Step 2 Arm A: LA ART vs Step 2 Arm B: SOC; The proportions of participants with HIV-1 RNA ≥ 200 copies/ml was compared by Fisher's Exact Test; Test type: Superiority; p < 0.001, Fisher Exact; Mean Difference (Final Values) = -24.5, 95% CI 2-sided [-36.1 to -12.8] — Difference in the proportions of participants with HIV-1 RNA ≥ 200 copies was calculated as LA-ART minus SOC

6. Secondary Outcome: Percentage of Participants With Plasma HIV-1 RNA Level Less Than 50 Copies/mL at Scheduled Study Visits on Steps 1
Description: Summarized the percentage of participants with plasma HIV-1 RNA level less than 50 copies/mL by study visit
Time Frame: Measured from Step 1 entry through Step 1, Week 20 visit
Population: Step 1 used Intention-to-Treat (ITT) population which was defined as all eligible participants who registered to Step 1, regardless of status on treatment.
Measure: Number; unit: percentage of participants
Groups:
- Step 1 SOC: In Step 1, All participants received SOC oral ART regimen for up to 24 weeks.
Arm/Group | Step 1 SOC
Number analyzed (Participants) | 453
percentage of participants
  Baseline | 21
  Week 4 | 57
  Week 8 | 47
  Week 12 | 55
  Week 16 | 56
  Week 20 | 63

7. Secondary Outcome: Percentage of Participants With Plasma HIV-1 RNA Level Less Than 200 Copies/mL at Scheduled Study Visits on Steps 1
Description: Summarized the percentage of participants with plasma HIV-1 RNA level less than 200 copies/mL by study visit
Time Frame: Measured from Step 1 entry through Step 1, Week 20 visit
Population: as for outcome 6
Measure: Number; unit: percentage of participants
Arm/Group | Step 1 SOC
Number analyzed (Participants) | 453
percentage of participants
  Baseline | 34
  Week 4 | 74
  Week 8 | 68
  Week 12 | 74
  Week 16 | 67
  Week 20 | 74

8. Secondary Outcome: Percentage of Participants With Plasma HIV-1 RNA Level Less Than 50 Copies/mL at Scheduled Study Visits on Steps 2
Description: Summarized the percentage of participants with plasma HIV-1 RNA level less than 50 copies/mL by study visit, and randomized treatment.
Time Frame: Measured from Step 2 entry through Step 2, Week 48 visit
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Step 2 Arm A: LA ART | Step 2 Arm B: SOC
Number analyzed (Participants) | 152 | 154
percentage of participants
  Baseline | 72 | 81
  Week 8 | 88 | 68
  Week 16 | 84 | 67
  Week 24 | 93 | 69
  Week 36 | 90 | 69
  Week 48 | 87 | 78

9. Secondary Outcome: Percentage of Participants With Plasma HIV-1 RNA Level Less Than 200 Copies/mL at Scheduled Study Visits on Steps 2
Description: Summarized the percentage of participants with plasma HIV-1 RNA level less than 200 copies/mL by study visit, and randomized treatment.
Time Frame: Measured from Step 2 entry through Step 2, Week 48 visit
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Step 2 Arm A: LA ART | Step 2 Arm B: SOC
Number analyzed (Participants) | 152 | 154
percentage of participants
  Baseline | 84 | 93
  Week 8 | 95 | 81
  Week 16 | 97 | 80
  Week 24 | 98 | 77
  Week 36 | 98 | 81
  Week 48 | 95 | 86

10. Secondary Outcome: Cumulative Probability of Discontinuation of Randomized Treatment in Step 2
Description: Permanent Step 2 treatment discontinuation was defined as premature discontinuation of randomized study treatment.
  Cumulative probability was calculated by Kaplan-Meier method.
Time Frame: Measured from Step 2 randomization through Step 2, Week 48 (up to 50 weeks)
Population: as for outcome 1
Measure: Number; unit: cumulative percent probability of event
Arm/Group | Step 2 Arm A: LA ART | Step 2 Arm B: SOC
Number analyzed (Participants) | 152 | 154
cumulative percent probability of event | 19.8 | 28.2
Statistical Analysis 1: Comparison: Step 2 Arm A: LA ART vs Step 2 Arm B: SOC; Treatment comparison was conducted by cumulative probability of permanent treatment discontinuation in Step 2 up to Step 2 Week 48 visit by treatment arm. The treatment difference was assessed using the 95% repeated confidence interval adjusted for interim efficacy analyses, i.e., a nominal 98.4% confidence interval; Test type: Superiority; Cumulative probability difference = -8.4, 98.4% CI 2-sided [-21.3 to 4.5] — Treatment difference in cumulative of permanent treatment discontinuation was calculated as LA-ART minus SOC.98.4% is nominal confidence interval

11. Secondary Outcome: Median Summary Score of HIV Treatment Satisfaction Questionnaire (HIVTSQ) in Step 2
Description: The questionnaire had 12 items rated using a 7-point Likert scale. Results were summarized as a total score that included 11 items, with the "pain/discomfort" item reported separately.
  1. The HIVTSQ "status" measured participant satisfaction with their current treatment with individual item rated ranging from 0 ("very dissatisfied") to 6 ("very satisfied") and the total score ranging from 0 to 66, where higher scores indicated a greater level of satisfaction with their HIV-1 treatment.
  2. The HIVTSQ "change" measured change in treatment satisfaction between a participant's previous and current treatment. The individual items were rated from -3 ("much less satisfied") to 3 ("much more satisfied") with a total score ranging from -33 to 33.
Time Frame: HIVTSQ status was collected on both arms at Step 2 entry and Week 24, and also at Week 48 for those randomized to SOC. At Week 48, HIVTSQ change was collected for participants on the LA-ART arm.
Population: Intention-to-Treat (ITT) Population was defined as all eligible participants who were randomized to the treatment arms, regardless of status on randomized treatment. Participants were assessed according to their randomized treatment, regardless of the treatment they received. Data were not collected from participants for HIVTSQ status for participants in LA-ART arm at week 24 or HIVTSQ change for participants in SOC arm at week 48
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Step 2 Arm A: LA ART | Step 2 Arm B: SOC
Number analyzed (Participants) | 152 | 154
score on a scale
  HIVTSQ status Week 0, 11-item total score | 63 [55 to 66] | 62 [53 to 66]
  HIVTSQ status Week 0, Satisfaction with pain/discomfort | 6 [5 to 6] | 6 [4 to 6]
  HIVTSQ status Week 24, 11-item total score | 66 [60 to 66] | 62 [51 to 66]
  HIVTSQ status Week 24, Satisfaction with pain/discomfort | 6 [5 to 6] | 6 [5 to 6]
  HIVTSQ status Week 48,11-item total score: number analyzed (Participants) | 0 | 154
  HIVTSQ status Week 48,11-item total score |  | 63 [51 to 66]
  HIVTSQ status Week 48, Satisfaction with pain/discomfort: number analyzed (Participants) | 0 | 154
  HIVTSQ status Week 48, Satisfaction with pain/discomfort |  | 6 [5 to 6]
  HIVTSQ change Week 24, 11-item total score | 0 [0 to 4] | 0 [0 to 1]
  HIVTSQ change Week 24, Satisfaction with pain/discomfort | 0 [0 to 0] | 0 [0 to 0]
  HIVTSQ change Week 48,11-item total score: number analyzed (Participants) | 152 | 0
  HIVTSQ change Week 48,11-item total score | 33 [31 to 33] |
  HIVTSQ change Week 48, Satisfaction with pain/discomfort: number analyzed (Participants) | 152 | 0
  HIVTSQ change Week 48, Satisfaction with pain/discomfort | 3 [2 to 3] |

12. Secondary Outcome: Number of Participants With Missed or Delayed Injections for Participants Who Received LA ART in Step 2
Description: Delayed injection was defined as 36-56 days from the previous injection. Missed injection was defined as the duration from the previous injection was longer than 56 days.
Time Frame: Measured from Step 2 randomization through Step 2, Week 52
Population: Analysis population was restricted to the participants who initiated injections
Measure: Number; unit: participants
Arm/Group | Step 2 Arm A: LA ART
Number analyzed (Participants) | 141
participants
  Delayed injection | 32
  Missed injection | 15

13. Secondary Outcome: Median of Summary Scores of HIV Treatment Adherence Self-Efficacy Scale in Step 1
Description: HIV Treatment Adherence Self-Efficacy Scale was a 12-item measure used to measure social and psychological determinants of adherence to ART among individuals living with HIV. The response scale to each individual item ranged from 0 ("cannot do at all") to 10 ("completely certain can do"). The total score reported was the average of all item scores, ranging from 0 to 10, with higher scores indicating higher adherence self-efficacy.
Time Frame: Step 1 entry, Weeks 12 and 20.
Population: as for outcome 6
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Step 1 SOC
Number analyzed (Participants) | 453
score on a scale
  Week 0 | 9 [7 to 10]
  Week 12 | 9 [7 to 10]
  Week 20 | 9 [8 to 10]

14. Secondary Outcome: Median of Summary Scores of HIV Treatment Adherence Self-Efficacy Scale in Step 2
Description: as for outcome 13
Time Frame: As Step 2 Week 0, Week 24 and Week 48
Population: As-treated Population was defined as all eligible participants who were randomized to the treatment arms and received at least one dose of a randomized treatment. Participants were assessed according to actual treatment strategy received.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Step 2 Arm A: LA ART | Step 2 Arm B: SOC
Number analyzed (Participants) | 151 | 152
score on a scale
  Week 0 | 9 [8 to 10] | 9 [8 to 10]
  Week 24 | 10 [8 to 10] | 10 [8 to 10]
  Week 48 | 10 [9 to 10] | 10 [8 to 10]

15. Secondary Outcome: Number of Participants With New Drug-resistance Mutations in Participants With Virologic Failure in Step 2
Description: Samples for HIV-1 resistance testing were collected at virologic failure confirmation visit. HIV-1 drug resistance mutations were determined using the IAS October/November 2022 Update of the Drug Resistance Mutations in HIV-1. New drug resistance mutations were defined as those detected at or after virologic failure which were not present at Step 1 screening/baseline.
  Virologic failure defined as two consecutive HIV-1 RNA > 200 copies/mL after Step 2 randomization, regardless of the time between them.
Time Frame: Measured at Step 1 screening/entry and at the time of virologic failure in Step 2
Population: Analysis population was restricted to the participants with virologic failure
Measure: Count of Participants; unit: Participants
Arm/Group | Step 2 Arm A: LA ART | Step 2 Arm B: SOC
Number analyzed (Participants) | 6 | 34
Participants
  With New Mutation | 2 | 2
  Without New Mutation | 3 | 20
  Discontinued study without a confirmation sample | 0 | 5
  Not done; HIV-1 RNA < 400 copies/mL | 1 | 4
  Sample Not Collected | 0 | 3

16. Secondary Outcome: Percentage of Participants With Grade 1 or Higher Injection Site Reactions (ISR) During Step 2
Description: Summarized and tabulated by number of participants with at least 1 injection site reactions.
  Severity Grade: 1 = Mild, 2 = Moderate, 3 = Severe, 4 = Life-Threatening, 5 = Death
Time Frame: Measured from Step 2 randomization through Step 2, Week 52
Population: Analysis population was restricted to participants who initiated injection
Measure: Number; unit: percentage of participant
Arm/Group | Step 2 Arm A: LA ART
Number analyzed (Participants) | 141
percentage of participant | 60

17. Secondary Outcome: Percentage of Participants Who Preferred Monthly Injections of Long-Acting HIV Treatment or Daily Oral HIV Treatment at Each Visit
Description: The Dichotomous Preference Questionnaire were:
  1. Monthly injections of Long-Acting HIV Treatment
  2. Daily oral HIV
Time Frame: Step 2 week 48, premature treatment visit, and study discontinuation visit
Population: Analysis population was restricted to the participants who had the indicated visit, either week 48, premature treatment discontinuation, or premature study discontinuation.
Measure: Number; unit: percentage of participants
Arm/Group | Step 2 Arm A: LA ART
Number analyzed (Participants) | 85
percentage of participants
  At Week 48, Daily oral HIV Treatment: number analyzed (Participants) | 78
  At Week 48, Daily oral HIV Treatment | 5
  At Week 48, Monthly injections of Long-Acting HIV Treatment: number analyzed (Participants) | 78
  At Week 48, Monthly injections of Long-Acting HIV Treatment | 95
  At Premature treatment discontinuation, Daily oral HIV Treatment: number analyzed (Participants) | 4
  At Premature treatment discontinuation, Daily oral HIV Treatment | 50
  At Premature treatment discontinuation, Monthly injections: number analyzed (Participants) | 4
  At Premature treatment discontinuation, Monthly injections | 50
  At Premature study discontinuation, Monthly injections: number analyzed (Participants) | 3
  At Premature study discontinuation, Monthly injections | 100

18. Secondary Outcome: Percentage of Participants With Opinions About Conditional Economic Incentive (CEI) Withdrawal
Description: The responses included: Not at all upset or disappointed, Not very upset or disappointed, Somewhat upset or disappointed, Extremely upset or disappointed, Undecided
Time Frame: At Step 2 entry and Step 2, Week 8
Population: Modified Intention-to-Treat (mITT) Population was defined as all eligible participants who were randomized to the treatment arms and received at least one dose of study treatment at or after randomization.
Measure: Number; unit: percentage of participants
Arm/Group | Step 2 Arm A: LA ART | Step 2 Arm B: SOC
Number analyzed (Participants) | 151 | 152
percentage of participants
  Week 0, Not at all upset or disappointed | 48 | 49
  Week 0, Not very upset or disappointed | 13 | 9
  Somewhat upset or Week 0, disappointed | 18 | 18
  Week 0, Extremely upset or disappointed | 11 | 11
  Week 0, Undecided | 9 | 14
  Week 8, Not at all upset or disappointed | 43 | 37
  Week 8, Not very upset or disappointed | 16 | 14
  Week 8, Somewhat upset or disappointed | 24 | 23
  Week 8, Extremely upset or disappointed | 12 | 17
  Week 8, Undecided | 5 | 10

19. Secondary Outcome: Median of Average Total Score of Step 1 HIV Treatment Adherence Self-Efficacy Scale Score (HIV-ASES)
Description: HIV-ASES was a 12-item measure used to measure social and psychological determinants of adherence to ART among individuals living with HIV. The response scale to each individual item ranged from 0 ("cannot do at all") to 10 ("completely certain can do"). The total score reported was the average of all item scores, ranging from 0 to 10, with higher scores indicating higher adherence self-efficacy.
Time Frame: Step 1 entry, Step 1 Weeks 12, and Step 1 Weeks 20
Population: as for outcome 6
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Step 1 SOC
Number analyzed (Participants) | 453
score on a scale
  Week 0 | 9 [7 to 10]
  Week 12 | 9 [7 to 10]
  Week 20 | 9 [8 to 10]

20. Secondary Outcome: Percentage of Participants With Missed Treatment Doses Among Participants Who Randomized to SOC Arm in Step 2
Description: The outcome was defined as participants with at least one dose missed in the last 30 days at each visit
Time Frame: At Step 2 entry, Step 2 week 4, Step 2 week 8, step 2 week 16, step 2 week 24, step 2 week 36, Step 2 week 48, and Step 2 week 52
Population: As-treated Population was defined as all eligible participants who were randomized to the treatment arms and received at least one dose of a randomized treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Step 2 ARM B: SOC
Number analyzed (Participants) | 152
percentage of participants
  Week 0 | 57
  Week 4 | 59
  Week 8 | 62
  Week 16 | 64
  Week 24 | 64
  Week 36 | 66
  Week 48 | 66
  Week 52 | 59

ADVERSE EVENTS:
Time Frame: From Step 1 entry to through Step 1, Week 24 and from Step 2 entry to through Step 2 Week 52 or premature study discontinuation. Summary of Adverse Events will be updated with Step 3 and 4 upon study completion.
Description: All grade ≥3, led to a change in study treatment/intervention regardless of grade, meeting SAE definition (as defined by ICH criteria) or EAE reporting requirement
  New diagnosis of diabetes or pre-existing diabetes with ≥Grade 2 diabetes,hepatitis B, hepatitis C, COVID-19 or SARS-CoV-2 infection, Cancer, Tuberculosis
  All ≥Grade 2 neurologic and psychiatric events, seizures regardless of grade
  Any bone fracture, ALT ≥3x ULN AND total bilirubin ≥2x ULN
Arm/Group | Step 1 SOC | Step 2 Arm A: LA-ART | Step 2 Arm B: SOC
All-Cause Mortality (participants affected / at risk) | 1/453 | 2/152 | 0/154
Serious Adverse Events (participants affected / at risk) | 38/453 | 21/152 | 16/154
Other Adverse Events (participants affected / at risk) | 73/453 | 40/152 | 37/154
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Step 1 SOC (N=453) | Step 2 Arm A: LA-ART (N=152) | Step 2 Arm B: SOC (N=154)
Acute left ventricular failure (Cardiac disorders) | 0 | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 2 | 0
Cardiac failure acute (Cardiac disorders) | 0 | 1 | 0
Coronary artery disease (Cardiac disorders) | 1 | 2 | 0
Left ventricular failure (Cardiac disorders) | 1 | 0 | 0
Photophobia (Eye disorders) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 2 | 0 | 1
Duodenitis (Gastrointestinal disorders) | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0
Peptic ulcer (Gastrointestinal disorders) | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 1
Alcoholic liver disease (Hepatobiliary disorders) | 0 | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0 | 0
Cirrhosis alcoholic (Hepatobiliary disorders) | 0 | 0 | 1
Abdominal sepsis (Infections and infestations) | 0 | 0 | 1
Abscess limb (Infections and infestations) | 0 | 0 | 2
Anal abscess (Infections and infestations) | 1 | 0 | 0
Appendicitis (Infections and infestations) | 1 | 0 | 0
Bronchitis viral (Infections and infestations) | 1 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 1
Cryptococcal fungaemia (Infections and infestations) | 1 | 0 | 0
Disseminated cryptococcosis (Infections and infestations) | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 2 | 0 | 0
Gastroenteritis shigella (Infections and infestations) | 0 | 1 | 0
Herpes zoster disseminated (Infections and infestations) | 0 | 0 | 1
Influenza (Infections and infestations) | 2 | 0 | 1
Mastitis (Infections and infestations) | 1 | 0 | 0
Neurosyphilis (Infections and infestations) | 1 | 0 | 0
Oesophageal candidiasis (Infections and infestations) | 1 | 0 | 0
Oropharyngeal candidiasis (Infections and infestations) | 0 | 0 | 1
Periumbilical abscess (Infections and infestations) | 0 | 0 | 1
Pharyngitis streptococcal (Infections and infestations) | 1 | 0 | 0
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 3 | 0 | 3
Pulmonary tuberculosis (Infections and infestations) | 0 | 0 | 1
Rotavirus infection (Infections and infestations) | 1 | 0 | 0
Sepsis (Infections and infestations) | 1 | 0 | 0
Shigella infection (Infections and infestations) | 0 | 1 | 0
Staphylococcal abscess (Infections and infestations) | 0 | 1 | 1
Superinfection bacterial (Infections and infestations) | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Gun shot wound (Injury, poisoning and procedural complications) | 1 | 0 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 1 | 1 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0
Blood bilirubin increased (Investigations) | 1 | 0 | 0
Haemoglobin decreased (Investigations) | 1 | 0 | 0
Abnormal loss of weight (Metabolism and nutrition disorders) | 1 | 0 | 0
Cachexia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Lactic acidosis (Metabolism and nutrition disorders) | 1 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
HER2 positive breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Ataxia (Nervous system disorders) | 0 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 2 | 1 | 0
Encephalopathy (Nervous system disorders) | 0 | 0 | 1
Headache (Nervous system disorders) | 1 | 0 | 0
Ischaemic cerebral infarction (Nervous system disorders) | 0 | 0 | 1
Metabolic encephalopathy (Nervous system disorders) | 0 | 1 | 0
Seizure (Nervous system disorders) | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0
Toxic encephalopathy (Nervous system disorders) | 0 | 1 | 0
Mixed anxiety and depressive disorder (Psychiatric disorders) | 0 | 1 | 0
Post-traumatic stress disorder (Psychiatric disorders) | 0 | 1 | 0
Psychotic disorder (Psychiatric disorders) | 0 | 1 | 0
Substance-induced psychotic disorder (Psychiatric disorders) | 1 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 1
Suicide attempt (Psychiatric disorders) | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 2 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Asthma late onset (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1
Lung perforation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Generalised bullous fixed drug eruption (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Neuropathic ulcer (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Substance use (Social circumstances) | 1 | 0 | 0
Drug therapy enhancement (Surgical and medical procedures) | 0 | 0 | 1
Hypotension (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Step 1 SOC (N=453) | Step 2 Arm A: LA-ART (N=152) | Step 2 Arm B: SOC (N=154)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0
Anogenital dysplasia (Gastrointestinal disorders) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 0 | 0
Food poisoning (Gastrointestinal disorders) | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 1 | 0
Vomiting (Gastrointestinal disorders) | 3 | 0 | 0
Chest pain (General disorders) | 1 | 0 | 0
Chills (General disorders) | 0 | 1 | 0
Facial discomfort (General disorders) | 0 | 1 | 0
Fatigue (General disorders) | 1 | 0 | 0
Injection site nodule (General disorders) | 0 | 2 | 0
Injection site pain (General disorders) | 0 | 5 | 0
Injection site swelling (General disorders) | 0 | 2 | 0
Peripheral swelling (General disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 1 | 1 | 0
Immune reconstitution inflammatory syndrome (Immune system disorders) | 1 | 0 | 0
Acute hepatitis C (Infections and infestations) | 0 | 1 | 0
Breakthrough COVID-19 (Infections and infestations) | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 1
COVID-19 (Infections and infestations) | 7 | 4 | 9
Cellulitis (Infections and infestations) | 1 | 0 | 0
Epstein-Barr virus infection (Infections and infestations) | 1 | 0 | 0
Hepatitis A (Infections and infestations) | 1 | 0 | 0
Joint abscess (Infections and infestations) | 1 | 0 | 0
Pelvic abscess (Infections and infestations) | 0 | 0 | 1
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 | 0 | 1
Pneumonia aspiration (Infections and infestations) | 0 | 1 | 0
Pneumonia respiratory syncytial viral (Infections and infestations) | 1 | 0 | 0
Suspected COVID-19 (Infections and infestations) | 0 | 1 | 0
Tonsillitis (Infections and infestations) | 0 | 1 | 0
Cartilage injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Incision site pain (Injury, poisoning and procedural complications) | 0 | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 1 | 1 | 0
Traumatic pain (Injury, poisoning and procedural complications) | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 3 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 2 | 2 | 1
Bilirubin conjugated increased (Investigations) | 2 | 0 | 0
Blood bilirubin increased (Investigations) | 2 | 0 | 0
Blood cholesterol increased (Investigations) | 0 | 1 | 1
Blood creatinine increased (Investigations) | 6 | 3 | 2
Blood glucose decreased (Investigations) | 0 | 1 | 0
Blood glucose increased (Investigations) | 2 | 3 | 2
Blood lactic acid increased (Investigations) | 0 | 1 | 0
Blood pressure increased (Investigations) | 1 | 1 | 1
Blood triglycerides increased (Investigations) | 1 | 1 | 0
Creatinine renal clearance decreased (Investigations) | 20 | 3 | 8
Creatinine renal clearance increased (Investigations) | 2 | 0 | 0
Glomerular filtration rate decreased (Investigations) | 1 | 0 | 0
Glycosylated haemoglobin increased (Investigations) | 1 | 0 | 0
Haemoglobin decreased (Investigations) | 1 | 1 | 1
Low density lipoprotein increased (Investigations) | 1 | 2 | 2
Neutrophil count decreased (Investigations) | 2 | 1 | 0
Platelet count decreased (Investigations) | 0 | 0 | 1
Abnormal loss of weight (Metabolism and nutrition disorders) | 3 | 1 | 0
Acidosis (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 2 | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 2 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Synovitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 0
Cervical radiculopathy (Nervous system disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 5 | 0 | 0
Hemiparesis (Nervous system disorders) | 0 | 1 | 0
Loss of consciousness (Nervous system disorders) | 0 | 1 | 0
Migraine (Nervous system disorders) | 1 | 0 | 0
Post herpetic neuralgia (Nervous system disorders) | 1 | 0 | 0
Seizure (Nervous system disorders) | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 2 | 0 | 1
Attention deficit hyperactivity disorder (Psychiatric disorders) | 1 | 0 | 0
Depressed mood (Psychiatric disorders) | 1 | 0 | 1
Depression (Psychiatric disorders) | 6 | 1 | 1
Drug abuse (Psychiatric disorders) | 0 | 1 | 0
Hypomania (Psychiatric disorders) | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 2 | 0 | 0
Mental status changes (Psychiatric disorders) | 0 | 0 | 1
Suicidal ideation (Psychiatric disorders) | 1 | 1 | 0
Diabetic nephropathy (Renal and urinary disorders) | 0 | 1 | 0
Glycosuria (Renal and urinary disorders) | 1 | 1 | 0
Nephropathy toxic (Renal and urinary disorders) | 1 | 0 | 0
Asthma late onset (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Hypertension (Vascular disorders) | 3 | 1 | 1

LIMITATIONS AND CAVEATS:
The trial was stopped per DSMB recommendation when the primary outcome measure did not meet the stopping criteria used at the interim efficacy review. Primary analysis included overrun data up to the DSMB review date and final confidence interval was adjusted for type I error spent at prior interim efficacy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In accordance with the Clinical Trials Agreement between NIAID (DAIDS) and company collaborators, NIAID (DAIDS) provides companies with a copy of any abstract, press release, or manuscript prior to submission for publication with sufficient time for company review and comment. The publication/other disclosure can be delayed for up to 30 additional business days for manuscripts and five (5) business days for abstracts, to preserve U.S. or foreign patent or other intellectual property rights.

DOCUMENTS (3):
  • Study Protocol and Informed Consent Form: Protocol Version 4.0 (2024-04-30): https://cdn.clinicaltrials.gov/large-docs/88/NCT03635788/Prot_ICF_000.pdf
  • Study Protocol and Informed Consent Form: Protocol Version 3.0 (2022-12-05): https://cdn.clinicaltrials.gov/large-docs/88/NCT03635788/Prot_ICF_001.pdf
  • Statistical Analysis Plan (2024-08-05): https://cdn.clinicaltrials.gov/large-docs/88/NCT03635788/SAP_002.pdf